CLINICAL TRIAL: NCT05691309
Title: Optimizing Vancomycin Therapy in Children
Acronym: Opt Vanc
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 22-020240; 5K23HD091365 (NIH)
Record Dates: First submitted 2022-12-29; First posted 2023-01-20 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Sepsis; Critical Illness; Infections; Drug Toxicity
MeSH Terms: conditions — Sepsis; Critical Illness; Infections; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Cohort: Recipients of vancomycin

SUMMARY:
The purpose of Opt Vanc is to evaluate the feasibility of Bayesian dose adaptation, based on a previously-developed population pharmacokinetic (PK) model and a single optimally timed PK sample, to predict vancomycin area under the curve (AUC) in critically ill children.

DETAILED DESCRIPTION:
Opt Vanc is an observational study of critically ill children prescribed IV vancomycin for a suspected infection at the Children's Hospital of Philadelphia. This study will evaluate how well Bayesian dose adaptation, based on a previously-developed population pharmacokinetic (PK) model for vancomycin and a single optimally timed vancomycin concentration, can predict vancomycin area under the curve (AUC) in critically ill children. Eligible subjects will be prescribed vancomycin and undergo routine therapeutic drug monitoring (TDM) per standard of care. At the time of TDM, each subject will have a vancomycin concentration obtained at the most informative sampling time to estimate AUC, as determined by the multiple-model optimal sampling function in PMetrics (population PK modeling program). Investigators will then compare the AUC determined using Bayesian estimation and the subject's optimally timed vancomycin concentration to the AUC determined using Bayesian estimation with all available concentrations (TDM samples plus the optimally timed sample). Investigators will also examine how AUC estimation compares to AUC calculated using standard-of-care methods (ie, log-linear equations). Further, Investigators will evaluate how well the population PK model, along with a subject's measured covariates and the optimally timed PK sample, can predict a subject's future vancomycin AUC.

ELIGIBILITY:
Inclusion Criteria:

* Administered intravenous vancomycin via intermittent infusion,
* Eligible for vancomycin AUC monitoring, per the subject's clinical team, and
* Parental/guardian permission (informed consent).

Exclusion Criteria:

* Receipt of renal replacement therapy, plasmapheresis, or extracorporeal membrane oxygenation (ECMO), or
* Unable to provide urine and blood samples.

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants aged 1-17 years receiving standard of care IV vancomycin for a suspected or confirmed infection will be enrolled at Children's Hospital of Philadelphia.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Downes KJ, Sharova A, Malone J, Odom John AR, Zuppa AF, Neely MN. Multiple Model Optimal Sampling Promotes Accurate Vancomycin Area-Under-the-Curve Estimation Using a Single Sample in Critically Ill Children. Ther Drug Monit. 2025 Jan 23;47(4):512-519. doi: 10.1097/FTD.0000000000001293. PMID 39846757

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on clinical receipt of IV vancomycin for a suspected infection and plans for therapeutic drug monitoring.
Pre-assignment Details: Of 29 enrolled participants, 22 met inclusion criteria and had optimal sampling time determination performed.
Period: Overall Study
Arm/Group | Study Cohort
Started | 22
Completed | 18
Not Completed | 4
Not completed — vancomycin discontinued by clinical team | 2
Not completed — vancomycin levels not evaluable | 2

BASELINE CHARACTERISTICS:
Population: Of 29 enrolled participants, 22 met inclusion criteria and had optimal sampling time determination performed.
Arm/Group | Study Cohort
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 6.1 [1.1 to 15.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 10
  More than one race | 0
  Unknown or Not Reported | 4
Weight [Median (Full Range); unit: kilograms] | 20 [9.5 to 73.2]
Estimated glomerular filtration rate (GFR) [Median (Full Range); unit: mL/min/1.73m^2] | 136 [40 to 178]

OUTCOME MEASURES:

1. Primary Outcome: 24-hour Vancomycin Area Under the Curve (AUC) From Optimally Timed Concentration
Description: This 24-hour vancomycin area under the curve (AUC) will be estimated using Bayesian estimation based on the population pharmacokinetic (PK) model, a subject's measured covariates and the optimally timed vancomycin concentration
Time Frame: within 24-48 hours following enrollment
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Study Cohort
Number analyzed (Participants) | 18
mg*hr/L | 494 [347 to 1008]

2. Secondary Outcome: 24-hour Vancomycin Area Under the Curve (AUC) Estimated Using All Available Vancomycin Concentrations
Description: This 24-hour vancomycin area under the curve (AUC) will be estimated using Bayesian estimation based on the population pharmacokinetic (PK) model, a subject's measured covariates and all available measured vancomycin concentrations
Time Frame: within 24-48 hours following enrollment
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Study Cohort
Number analyzed (Participants) | 18
mg*hr/L | 495 [336 to 1084]

3. Secondary Outcome: 24-hour Vancomycin Area Under the Curve (AUC) Calculated Using Standard-of-care Methods
Description: This 24-hour vancomycin area under the curve (AUC) will be calculated using standard clinical methods (Zaske-Sawchuk method)
Time Frame: within 24-48 hours following enrollment
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Study Cohort
Number analyzed (Participants) | 18
mg*hr/L | 526 [258 to 1111]

4. Secondary Outcome: Visit 2 Vancomycin Area Under the Curve (AUC) Using Optimally Timed Concentration
Description: The predicted 24-hour vancomycin area under the curve (AUC) at visit 2 will be estimated using Bayesian estimation based on the population pharmacokinetic (PK) model, a subject's measured covariates and the optimally timed vancomycin concentration at visit 1
Time Frame: 24-72 hours after visit 1
Population: Given the short timeframe, only 11 subjects had data available for this outcome measure.
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Study Cohort
Number analyzed (Participants) | 11
mg*hr/L | 500 [326 to 668]

5. Secondary Outcome: Visit 2 Vancomycin Area Under the Curve (AUC) Using All Available Vancomycin Concentrations
Description: The predicted 24-hour vancomycin area under the curve (AUC) at visit 2 will be estimated using Bayesian estimation based on the population pharmacokinetic (PK) model, a subject's measured covariates and all available vancomycin concentrations
Time Frame: 24-72 hours after visit 1
Population: Given the short timeframe, only 11 subjects had data available for this outcome measure.
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Study Cohort
Number analyzed (Participants) | 11
mg*hr/L | 502 [370 to 681]

6. Secondary Outcome: Visit 2 Vancomycin Area Under the Curve (AUC) Calculated Using Standard-of-care Methods
Description: This 24-hour vancomycin area under the curve (AUC) will be calculated using standard clinical methods (Zaske-Sawchuk method) based on measured concentrations at visit 2
Time Frame: 24-72 hours after visit 1
Population: Given the short timeframe, only 7 subjects had data available for this outcome measure.
Measure: Median (Full Range); unit: mg*hr/L
Arm/Group | Study Cohort
Number analyzed (Participants) | 7
mg*hr/L | 486 [305 to 754]

ADVERSE EVENTS:
Description: Adverse Events were not monitored/assessed as this was an observational study.
Arm/Group | Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT05691309/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/09/NCT05691309/ICF_001.pdf